CLINICAL TRIAL: NCT00391963
Title: Comparison of the Bispectral Index and the Entropy of the Electroencephalogram During Total Intravenous Anesthesia
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Other Study IDs: Foch-2
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Bispectral index, Entropy

SUMMARY:
To compare Bispectral index and entropy during maintenance of anesthesia

DETAILED DESCRIPTION:
Several monitors are currently proposed to evaluate the depth of hypnosis. Among them, Bispectral Index (BIS) is a well known and widely used parameter derived from the patient's electroencephalograph (EEG). Spectral entropy relies on the extent of disorder in both EEG and electromyography (EMG) signals and returns 2 values: State Entropy (SE) and Response Entropy. SE is computed over the frequency range of 0.8-32 Hz and reflects the level of hypnosis while Response Entropy is computed over the frequency range of 0.8-47 Hz and reflects also EMG activity. BIS and SE are dimensionless numbers scaled from 100 to 0 for BIS and from 91 to 0 for SE.

The BIS and Entropy manufacturers claim that adequate level of anesthesia is defined by a BIS or SE value between 40 and 60. But some observations have shown that the monitors provided different information. These observations led us to carry out this prospective observational study designed to study the comparability between BIS and SE during the maintenance period of propofol-sufentanil anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* American Society of Anesthesiologists physical status 1-3,
* surgery under general anesthesia using propofol, sufentanil, and a relaxant agent,
* surgery lasting more than one hour,
* tracheal extubation planned at end of surgery

Exclusion Criteria:

* pregnant women,
* allergy to propofol,
* neurological or muscular disorder,
* treatment with opioids or any psychoactive medication,
* cardiac surgery,
* thyroid disorder,
* emergency surgery,
* prone or lateral decubitus position (difficulty to have a correct probe position)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2006-06; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Principal Investigator — Hôpital Foch
Locations (2):
- France (2):
  - Dept of Anesthesia and Intensive Care, Hôpital Beaujon, Clichy
  - Dept of Anesthesiology, Hôpital Foch, Suresnes

REFERENCES:
- [Background] Schmidt GN, Bischoff P, Standl T, Hellstern A, Teuber O, Schulte Esch J. Comparative evaluation of the Datex-Ohmeda S/5 Entropy Module and the Bispectral Index monitor during propofol-remifentanil anesthesia. Anesthesiology. 2004 Dec;101(6):1283-90. doi: 10.1097/00000542-200412000-00007. PMID 15564934
- [Background] Vanluchene AL, Vereecke H, Thas O, Mortier EP, Shafer SL, Struys MM. Spectral entropy as an electroencephalographic measure of anesthetic drug effect: a comparison with bispectral index and processed midlatency auditory evoked response. Anesthesiology. 2004 Jul;101(1):34-42. doi: 10.1097/00000542-200407000-00008. PMID 15220769
- [Derived] Aime I, Gayat E, Fermanian C, Cook F, Peuch C, Laloe PA, Mantz J, Fischler M. Effect of age on the comparability of bispectral and state entropy indices during the maintenance of propofol-sufentanil anaesthesia. Br J Anaesth. 2012 Apr;108(4):638-43. doi: 10.1093/bja/aer457. Epub 2012 Jan 17. PMID 22258203